CLINICAL TRIAL: NCT06628609
Title: Post-exercise Therapeutic Modalities on Functional Performance, Muscle Damage and Oxidative Stress of CrossFit® Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full Professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3.997.120
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Exercise Recovery
Keywords: Therapeutic modalities; Exercise recovery; Muscle damage; Oxidative stress
MeSH Terms: interventions — Extracorporeal Shockwave Therapy; Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Control (Other): Passive recovery for 30 minutes
  Interventions: Other: Passive recovery
- PBMT-sMF (Experimental): Photobiomodulation therapy combined with static magnetic field, with a total treatment duration lasting for around 30 minutes.
  Interventions: Device: PBMT-sMF
- Shock wave (Active Comparator): Shock wave therapy applied for 30 minutes.
  Interventions: Device: Shock wave
- Pneumatic compression (Active Comparator): Pneumatic compression applied for 30 minutes.
  Interventions: Device: Pneumatic compression

INTERVENTIONS:
Other: Passive recovery — Volunteers laid in supine position resting for 30 minutes.
  Arms: Control
Device: PBMT-sMF — PBMT-sMF applied in the lower limbs with different doses per muscle group.
  Arms: PBMT-sMF
Device: Shock wave — Shock wave therapy applied in the lower limbs for 30 minutes.
  Arms: Shock wave
Device: Pneumatic compression — Pneumatic compression applied in the lower limbs for 30 minutes.
  Arms: Pneumatic compression

SUMMARY:
Crossfit® is a training modality that consists in functional movements, constantly varied and executed at high intensity. Both training sessions and competitions involve physically demanding activities, which in addition to being performed at very high intensity also involves the aerobic metabolism pathway. These characteristics led to very high metabolic and muscular stress, as well as decrease in physical performance immediately after competitions and training sessions. The cumulative effects of the metabolic and muscular stress can be a precursor of injuries. Studies using different therapeutic modalities aiming to improve post-exercise recovery are needed in order to tackle this issue.

Oxidative stress induced by exercise has been a research field in constant growth, due to its relationship with the processes of fatigue, decreased production of muscle strength, and its ability to cause damage to the cell.

To the date there are no studies comparing the effects of different therapeutic modalities applied after an exercise session on functional performance, muscle damage, and oxidative stress in an exercise modality such as Crossfit®.

Therefore, the aim of this project is to assess and compare the effects of different therapeutic modalities on functional performance, muscle damage, and oxidative stress of Crossfit® athletes.

DETAILED DESCRIPTION:
A randomized, crossover, controlled trial will be carried out.

All volunteers will be allocated to four interventions, and the order of the interventions will be randomized.

The outcomes will be assessed at baseline (prior to the Workout of the Day - WOD), and in different timepoints after the WOD.

The WOD will be consisted in finishing as quickly as possible a sequence of three exercises (Calories in Assault AirBike®, Hang Squat Clean and Box Jump Over), in a well-known series model for the athletes, without rest.

The investigators will analyze functional performance, biochemical markers of muscle damage and oxidative stress, the ratings of perceived exertion, and the volunteers satisfaction with the interventions.

All data will be analyzed both in their absolute values and in relation to their percentage variation from the values obtained in the pre-WOD (baseline) assessments.

ELIGIBILITY:
Inclusion Criteria: - Crossfit® amateur male athletes; - Do not present a history of musculoskeletal injury in the regions of the hips, knees and calves in the month preceding the study; - Are not using pharmacological agents; - Athletes should have been practicing the sport for at least 1 year; - Voluntarily commit to participate in all stages of the study.

Exclusion Criteria: - Present musculoskeletal or joint injuries during data collection; - Present history of musculoskeletal injury in the regions of the hips, knees and calves in the month preceding the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender men.
Enrollment: 12 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-11-03 (Actual); Study Completion 2024-11-03 (Actual)

PRIMARY OUTCOMES:
Change in functional performance | 1 hour after WOD (workout of the day).
  The functional performance will be assessed through the countermovement jump (CMJ) test.

SECONDARY OUTCOMES:
Change in functional performance | 24 hours and 48 hours after WOD (workout of the day)
  The functional performance will be assessed through the countermovement jump (CMJ) test.
Change in the activity of lactate dehydrogenase (LDH) | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  The activity of LDH will be analyzed from the blood samples collected from the participants through spectrophotometry and using specific reagent kits.
Change in thiobarbituric acid (TBARS) | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  TBARS will be analyzed from the blood samples collected from the participants through spectrophotometry and using specific reagent kits.
Change in carbonylated proteins | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  Carbonylated proteins will be analyzed from the blood samples collected from the participants through spectrophotometry and using specific reagent kits.
Change in catalase (CAT) activity | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  CAT activity will be analyzed from the blood samples collected from the participants through spectrophotometry and using specific reagent kits.
Change in superoxide dismutase (SOD) activity | 1 hour, 24 hours and 48 hours after WOD (workout of the day).
  SOD activity will be analyzed from the blood samples collected from the participants through spectrophotometry and using specific reagent kits.
Participants' perceived exercise intensity | 1 minute after WOD (workout of the day), 1 minute post-treatment/intervention, 1 hour, 24 hours and 48 hours after WOD.
  The perception of exercise intensity will be assessed through a 0-100 Ratings of Perceived Exertion Scale: in this scale lower score, means lower degree of fatigue and higher score, means higher degree of fatigue.
Participants' satisfaction regarding the interventions | 48 hours after WOD (workout of the day).
  The participants satisfaction regarding the interventions will be assessed through the LIKERT scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Pinto Leal Junior, Ph.D., M.Sc., PT., Principal Investigator — Nove de Julho University
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon request addressed to the principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available six months after the manuscript publication for five years after that.
Access Criteria: All IPD that underlie results in a publication will be available on reasonable request.